CLINICAL TRIAL: NCT01618227
Title: A Prospective Randomized Trial of Rehabilitation With or Without Static Progressive Splinting for Wrist Stiffness
Brief Title: Rehabilitation With or Without Static Progressive Splinting for Wrist Stiffness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a lack of resources and the principal investigator leaving the institution, we stopped the study prior to reaching enrollment target.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007P002509
Record Dates: First submitted 2012-06-07; First posted 2012-06-13 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-02

CONDITIONS: Post-traumatic Stiff Wrists
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation with static progressive splinting (Experimental): Static progressive splinting is a well-established adjunct for restoring motion in stiff joints. Such splints apply a static stress relaxation force to the wrist and forearm tissues, which is sequentially increased as motion is achieved.
  Interventions: Device: Joint Active Systems (JAS) Static progressive splint
- Rehabilitation without splinting (Experimental)
  Interventions: Procedure: Rehabilitation without splinting

INTERVENTIONS:
Device: Joint Active Systems (JAS) Static progressive splint — Subjects will have a standard rehabilitation program including physical or occupational therapy and home exercises throughout the study. Upon receipt of the splint, subjects will be instructed in proper application and use by their treating therapist or a representative of the company. Subjects will be instructed to follow the daily splint wearing protocol provided by the device manufacturer.
  Arms: Rehabilitation with static progressive splinting
Procedure: Rehabilitation without splinting — Subjects will have a standard rehabilitation program including physical or occupational therapy and home exercises without additional splinting.
  Arms: Rehabilitation without splinting

SUMMARY:
Loss of wrist flexion and extension is a common problem after wrist and forearm fractures that may lead to disability and unsatisfactory outcomes after fracture treatment. In many patients, this range of motion loss is caused by stiffness of the soft tissues. Such stiffness may loosen up and improve with rehabilitation. Static progressive splints apply a constant stretch upon the wrist resulting in a stretch relaxation and plastic deformation of the soft tissues. By altering the splint's bending angle, one can incrementally increase the force applied on either wrist flexion or extension. There are no data comparing rehabilitation with static-progressive splinting to rehabilitation without static-progressive splinting for the restoration of wrist flexion and extension after wrist or forearm fractures.

Primary study hypothesis:

Two months after study enrollment patients that use static progressive splinting have better wrist flexion and extension than patients that use standard therapy techniques.

Secondary study hypotheses:

1. Six months after study enrollment, subjects that use static progressive splinting have better wrist flexion and extension than those that use standard therapy techniques.
2. Motion at enrollment, 2 months and 6 months after enrollment correlates with negative pain thoughts, pain anxiety, and depression.
3. Six months after study enrollment, subjects that use static progressive splinting have had fewer physical/occupational therapy visits than those that use standard therapy techniques.
4. Six months after study enrollment patients that use static progressive splinting have had fewer additional surgeries than patients that use standard therapy techniques.

This study will employ a prospective randomized design. Subjects will be invited to enroll during their routine office follow-up visit. Informed consent will be obtained. Subjects will be randomized on a 1:1 ratio to rehabilitation with or without static progressive splinting.

All subjects will have a standard rehabilitation program including physical or occupational therapy and home exercises throughout the study. The static progressive splint will be prescribed according to the randomization sequence. Upon receipt of the splint, subjects will be instructed in proper application and use by their treating therapist or a representative of the company. Subjects will be instructed to follow the daily splint wearing protocol provided by the device manufacturer. Use of the splints will be discontinued at the patient's discretion or when a plateau phase in active range of motion is achieved (defined as no measurable gains in active range of motion achieved in a 30-day period).

DETAILED DESCRIPTION:
Upon enrollment, a form containing demographic and injury-related information will be completed, and the subjects will fill out the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire. Subjects will be evaluated for negative pain thoughts, pain anxiety, and depression. Study staff will supervise and assist with the questionnaires. Subjects will be evaluated at 2 and 6 months after enrollment during their routine office visits. The DASH questionnaire will be filled out and active wrist motion will be measured using a standard goniometer by a research assistant who will not be involved in the care of the patient. The number of physical/occupational therapy visits, additional surgeries, ease of splint application and use, and splint protocol compliance will be recorded.

The investigators intend to study the effectiveness rather than the efficacy of the splint, which means subjects will be free at all times to pursue an alternative treatment course and discontinue splint wear. The investigators will use intention to treat analysis.

Radiographs and other diagnostic studies will be obtained at the discretion of the treating surgeon and will not differ from routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Less than 45 degrees of wrist extension, flexion, or both.
* Between two weeks and six months after a wrist or forearm fracture

Exclusion Criteria:

* Active infection
* Wound problems
* Inability to comply with a structured rehabilitation protocol
* Burn-related contractures
* Primary osteoarthritis
* Clinically significant anatomic deformity, implants, or heterotopic bone hindering motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rehabilitation With Static Progressive Splinting | Rehabilitation Without Splinting
Started | 2 | 2
Completed | 2 | 0
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rehabilitation With Static Progressive Splinting | Rehabilitation Without Splinting | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (3.5) | 53.5 (3.9) | 55 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Wrist Range of Motion
Description: Flexion and extension of the wrist will be measured with a goniometer in degrees, the sum of which will determine range of motion.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rehabilitation With Static Progressive Splinting | Rehabilitation Without Splinting
Number analyzed (Participants) | 2 | 2
degrees | 36.5 (9.19) | 57.5 (10.6)

2. Secondary Outcome: Wrist Range of Motion
Description: as for outcome 1
Time Frame: 6 months
Population: Two subjects had the same range of motion at 6 months, therefore SD is 0.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rehabilitation With Static Progressive Splinting | Rehabilitation Without Splinting
Number analyzed (Participants) | 2 | 0
degrees | 45 (0) |

3. Secondary Outcome: Number of Physical/Occupational Therapy Visits
Description: Number of physical/occupational therapy visits will be collected from enrollment.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Rehabilitation With Static Progressive Splinting | Rehabilitation Without Splinting
Number analyzed (Participants) | 2 | 0
visits | 28 (5.66) |

4. Secondary Outcome: Number of Additional Surgeries
Description: The number of additional surgeries will be recorded and compared between groups.
Time Frame: 6 months
Measure: Number; unit: Number of Additional Surgeries
Arm/Group | Rehabilitation With Static Progressive Splinting | Rehabilitation Without Splinting
Number analyzed (Participants) | 2 | 0
Number of Additional Surgeries | 0 |

ADVERSE EVENTS:
Arm/Group | Rehabilitation With Static Progressive Splinting | Rehabilitation Without Splinting
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No